CLINICAL TRIAL: NCT04133857
Title: Acute Effects of High Intensity Interval Training (HIIT) and Steady State Moderate Intensity Training (SSMIT) on Intraocular Pressure Among Sedentary Individuals
Brief Title: Acute Effects of HIIT and SSMIT on Intraocular Pressure Among Sedentary Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Prof Mohd Nahar Azmi Mohamed, associate professor, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20171031-5738
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): undergo HIIT first then SSMIT protocol
  Interventions: Other: aerobic exercise
- Group B (Active Comparator): undergo SSMIT first then HIIT protocol
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — aerobic exercise HIIT : High intensity interval training SSMIT : Steady state moderate intensity training

SUMMARY:
Purpose to study the acute effects of both forms of aerobic exercise (HIIT and SSMIT) on intraocular pressure among healthy sedentary individuals

DETAILED DESCRIPTION:
40 participants were recruited and divided into 2 groups. Each group performed 2 exercise protocols with a 4 day washout period between them.

The intraocular pressure was measured before the exercise and after the exercise in 5 minute periods up until 30 minutes post exercise.

The intraocular pressure was measured using a handheld rebound tonometer.

ELIGIBILITY:
Inclusion Criteria:

* all University hospital staff

Exclusion Criteria:

* previous ocular trauma
* surgery in the eligible eye
* known case of glaucoma or glaucoma suspect (IOP > 21mmHg)
* history of glaucoma laser procedure/surgery within 6 months in eligible eye
* unable to undergo IOP measurements
* undiagnosed visual condition
* any uncontrolled medical condition such as end stage renal failure, uncontrolled diabetes and uncontrolled hypertension

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure | 30 minutes
  changes in intraocular pressure before and after exervcise

SECONDARY OUTCOMES:
compare which form of exercise (HIIT & SSMIT) is superior in reducing intraocular pressure | 30 days
  difference in intraocular pressure reduction observed between each exercise protocol

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya, Kuala Lumpur, Wilayah Perseketuan, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04133857/Prot_SAP_000.pdf